CLINICAL TRIAL: NCT03217058
Title: Implementing Computerized Substance Use and Depression Screening and Evidence-based Treatments in an HIV Primary Care Population
Brief Title: Computerized Substance Use and Depression Screening and Behavioral Treatment in HIV Primary Care
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-20272; K24AA025703 (NIH); R01DA043139 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorders; HIV; Depression; Anxiety
Keywords: digital health; implementation; primary care
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design evaluating implementation of computerized screening and behavioral interventions delivered by primary care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation (No Intervention): The pre-implementation cohort includes data from 5000 HIV primary care clinic patients in Kaiser Permanente Northern California, who receive services prior to implementation of computerized screening and behavioral intervention in the clinics.
- Post-implementation (Experimental): The post-implementation cohort includes data from 5000 HIV primary care clinic patients in Kaiser Permanente Northern California, who receive services after computerized screening and behavioral intervention have been implemented in the clinics.
  Interventions: Behavioral: Clinic-based screening and behavioral interventions

INTERVENTIONS:
Behavioral: Clinic-based screening and behavioral interventions — As part of routine HIV primary care visits, patients will complete self-administered computerized substance use, anxiety and depression screening measures. Results will be integrated into the electronic health record. A behavioral health specialist on the clinic staff will contact patients who screen positive for high-risk substance use, anxiety or depression, and offer behavioral interventions including motivational interviewing and cognitive behavioral therapy.
  Arms: Post-implementation

SUMMARY:
Substance use disorders (SUDs), depression and anxiety in HIV-infected patients result in poor HIV outcomes, yet are often unrecognized and untreated. To address these problems, this study examines the implementation and effectiveness of a clinical intervention consisting of self-administered tablet-based SUD and depression screening at routine HIV primary care clinic visits, followed by evidence-based treatments for SUD, anxiety and depression delivered by a behavioral health specialist. If successful, this study has potential to reduce SUD-, anxiety- and depression-related problems and reduce HIV treatment disparities for patients with these comorbidities.

DETAILED DESCRIPTION:
Substance use disorders (SUDs), anxiety and depression are common among HIV-positive patients and lead to poor HIV treatment outcomes and increased mortality. Yet these disorders often go unrecognized and untreated, despite the availability of effective interventions. To enhance HIV care, this study examines the impact of self-administered tablet-based screening for SUD risk, anxiety and depression using validated measures, with results integrated into the electronic health record and reviewed by behavioral health specialists (BHSs) embedded in primary care HIV clinics. Based on screening results, BHSs will initiate motivational interviewing (MI)- and cognitive behavioral therapy (CBT)-based clinical interventions. Using a hybrid study approach, the investigators will evaluate both implementation and effectiveness of screening and intervention. Specifically, the investigators will employ a stepped-wedge trial design, with a 12-month intervention phase implemented sequentially in the 3 largest HIV primary care clinics serving 5000 HIV-positive patients in Kaiser Permanente Northern California (KPNC), with a 12-month usual care period prior to implementation in each clinic functioning as an observational phase for comparison. This design, a variation of a cross-over RCT, allows for intervention refinement at each clinic and provides the opportunity to compare outcomes among patients before and after implementation. The investigators will evaluate patient-level (e.g., demographics, HIV, SUD, anxiety and depression severity) and provider-level (e.g., provider attitudes) factors affecting implementation and effectiveness, and will analyze cost effectiveness. The results of the study will provide insights regarding the implementation of evidence-based treatments for SUD, anxiety and depression, such as: 1) How self-administered computerized SUD, anxiety and depression screening and corresponding behavioral interventions can be effectively and efficiently implemented in HIV primary care clinics and sustained over time; 2) What patient and clinic characteristics influence screening and intervention rates; 3) To what extent implementation of screening and treatment impacts SUD and depression outcomes, as well as HIV outcomes, including retention in care, viral suppression and Veterans Aging Cohort Study index score, and 4) What are the barriers, facilitators and costs of implementation. The study setting is generalizable to other HIV clinics and health systems and will provide key data regarding the effective delivery of treatment options within primary care settings, and in coordination with SUD and psychiatry specialty care. Furthermore, the study addresses NIH-identified high priority HIV research topics since effective treatment of SUDs and/or depression anxiety would alleviate HIV treatment disparities for these individuals and reduce SUD-, anxiety and depression-related medical comorbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adults

Exclusion Criteria:

* Patients under age 18

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10821 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Satre, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lea AN, Levine TM, Davy-Mendez T, Leibowitz A, Altschuler A, Flamm J, Hare CB, N Luu M, Silverberg MJ, Satre DD. Mental health and substance use screening in HIV primary care before and during the early COVID-19 pandemic. BMC Health Serv Res. 2023 May 16;23(1):494. doi: 10.1186/s12913-023-09477-6. PMID 37194051
- [Derived] Lea AN, Altschuler A, Leibowitz AS, Levine-Hall T, McNeely J, Silverberg MJ, Satre DD. Patient and provider perspectives on self-administered electronic substance use and mental health screening in HIV primary care. Addict Sci Clin Pract. 2022 Feb 9;17(1):10. doi: 10.1186/s13722-022-00293-7. PMID 35139911
- [Derived] Satre DD, Anderson AN, Leibowitz AS, Levine-Hall T, Slome S, Flamm J, Hare CB, McNeely J, Weisner CM, Horberg MA, Volberding P, Silverberg MJ. Implementing electronic substance use disorder and depression and anxiety screening and behavioral interventions in primary care clinics serving people with HIV: Protocol for the Promoting Access to Care Engagement (PACE) trial. Contemp Clin Trials. 2019 Sep;84:105833. doi: 10.1016/j.cct.2019.105833. Epub 2019 Aug 22. PMID 31446142

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intervention was implemented sequentially at three clinics, starting in Oakland on 10/30/2018, next in Sacramento on 2/1/2019 and finally on 6/1/2019 in San Francisco, and continued until 7/17/2020 in all 3 clinics. In each clinic an observation period of 12 to 24 months prior to implementation was designated as pre-intervention period, depending on the analyses. Analyses were done at the participant level, not at the clinic level, and compared pre- and post-implementation periods.
Groups:
- Oakland Clinic: HIV positive participants who received primary care at the Oakland clinic
- Sacramento Clinic: HIV positive participants who received primary care at the Sacramento clinic
- San Francisco Clinic: HIV positive participants who received primary care at the San Francisco clinic
Period: Pre-Implementation
Arm/Group | Oakland Clinic | Sacramento Clinic | San Francisco Clinic
Started | 1507 | 1011 | 3188
Completed | 1507 | 1011 | 3188
Not Completed | 0 | 0 | 0
Period: Post-Implementation
Arm/Group | Oakland Clinic | Sacramento Clinic | San Francisco Clinic
Started | 1528 | 986 | 2601
Completed | 1528 | 986 | 2601
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-implementation | Post-implementation | Total
Number analyzed (Participants) | 5706 | 5115 | 10821
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 3 | 9
  Between 18 and 65 years | 5034 | 4335 | 9369
  >=65 years | 666 | 777 | 1443
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 418 | 425 | 843
  Male | 5288 | 4690 | 9978
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 27 | 55
  Asian | 374 | 332 | 706
  Native Hawaiian or Other Pacific Islander | 25 | 24 | 49
  Black or African American | 1022 | 993 | 2015
  White | 3123 | 2680 | 5803
  More than one race | 180 | 157 | 337
  Unknown or Not Reported | 954 | 902 | 1856
Region of Enrollment [Number; unit: participants]
  United States | 5706 | 5115 | 10821
Study Clinic [Number; unit: participants]
  Oakland | 1507 | 1528 | 3035
  Sacramento | 1011 | 986 | 1997
  San Francisco | 3188 | 2601 | 5789
HIV Transmission Risk factor [Number; unit: participants]
  MSM | 4337 | 3834 | 8171
  Heterosexual | 600 | 601 | 1201
  IDU | 408 | 363 | 771
  Other/Unknown | 361 | 317 | 678
CD4 cells [Number; unit: participants]
  <200 T cells/ul | 193 | 198 | 391
  200-350 T cells/ul | 373 | 378 | 751
  350-500 T cells/ul | 657 | 662 | 1319
  >500 T cells/ul | 3308 | 2900 | 6208
  No lab results in prior 365 days | 1175 | 977 | 2152
Viral load [Number; unit: participants]
  <200 copies/mL | 4754 | 4356 | 9110
  >=200 copies/mL | 409 | 341 | 750
  No lab results in prior 365 days | 543 | 418 | 961

OUTCOME MEASURES:

1. Primary Outcome: Change in Mental Health and Substance Use Screening Rates
Description: Rate of screening using usual care methods (pre-implementation) compared with rate of screening using computerized methods, based on electronic health record (EHR) data.
Time Frame: 12 months pre-implementation period to the end of the implementation period, up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation | Post-implementation
Number analyzed (Participants) | 5706 | 5115
Participants | 2008 | 2379

2. Primary Outcome: Treatment Rate
Description: Initiation of substance use, anxiety and depression treatment services, based on EHR data
Time Frame: Percent treated by 6 months after newly identified substance use
Measure: Count of Participants; unit: Participants
Groups:
- Post-implementation (Clinical); Post-implementation (Survey): The post-implementation cohort includes data from 5000 HIV primary care clinic patients in Kaiser Permanente Northern California, who receive services after computerized screening and behavioral intervention have been implemented in the clinics.
  Clinic-based screening and behavioral interventions: As part of routine HIV primary care visits, patients will complete self-administered computerized substance use, anxiety and depression screening measures. Results will be integrated into the electronic health record. A behavioral health specialist on the clinic staff will contact patients who screen positive for high-risk substance use, anxiety or depression, and offer behavioral interventions including motivational interviewing and cognitive behavioral therapy.
Arm/Group | Pre-implementation | Post-implementation (Clinical) | Post-implementation (Survey)
Number analyzed (Participants) | 1135 | 238 | 746
Participants
  Any treatment | 375 | 83 | 194
  Medication Only | 261 | 50 | 127
  BHS only | 136 | 26 | 75
  Specialty Care Only | 91 | 24 | 22

3. Primary Outcome: Treatment Rate
Description: Initiation of substance use, anxiety and depression treatment services, based on EHR data
Time Frame: Percent treated by 6 months after newly identified mental health problem
Measure: Number; unit: participants
Arm/Group | Pre-implementation | Post-implementation (Clinical) | Post-implementation (Survey)
Number analyzed (Participants) | 1300 | 341 | 347
participants
  Any treatment | 1079 | 249 | 226
  Medication Only | 962 | 228 | 191
  BHS only | 221 | 44 | 49
  Specialty Care Only | 455 | 95 | 90

4. Secondary Outcome: Change in Substance Use Severity: Tobacco, Alcohol, Prescription Medication, and Other Substance Use Tool (TAPS)
Description: Unadjusted mean change of screening scores for Tobacco, alcohol, and cannabis use from first post intervention screen to second post intervention screen using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) tool. The score ranges from zero - 3 for each substance, zero indicating no use and 2 or higher indicating high-risk, for each substance. 0 = No Use in Past 3 Months, 1 = Problem Use, and 2+ = Higher Risk.
Time Frame: First post intervention screen (1 month) to second post intervention screen (21 months)
Population: Of 2,865 people with HIV screened across all three clinics post-intervention, 403 screened positive at first screen AND completed a follow-up screen.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Change in Post-intervention Positive Substance Use Screens: Change in post-intervention positive substance use screens between first post-intervention substance use screen and second post-intervention substance use screen
Arm/Group | Change in Post-intervention Positive Substance Use Screens
Number analyzed (Participants) | 403
scores on a scale
  Tobacco | -0.36 [-0.49 to -0.23]
  Alcohol | -0.72 [-0.87 to -0.58]
  Cannabis | -0.61 [-0.75 to -0.47]

5. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder 2-item (GAD-2) Scores
Description: Unadjusted mean change of screening scores for depression and anxiety from first post intervention screen to second post intervention screen.
  The PHQ-9 assesses degree of depression severity. The score ranges from zero - 27 with higher scores indicate higher depression.
  GAD-2 assesses degree of anxiety severity. The score ranges from zero - 6 with higher scores indicate higher anxiety.
Time Frame: First post intervention screen (1 month) to second post intervention screen (21 months)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Change in Post-intervention Positive Depression and Anxiety Screens: Change in post-intervention positive depression and anxiety screens between first post-intervention depression or anxiety screen and second post-intervention depression or anxiety screen
Arm/Group | Change in Post-intervention Positive Depression and Anxiety Screens
Number analyzed (Participants) | 403
scores on a scale
  Depression (GAD-2) | -5.25 [-6.44 to -4.06]
  Anxiety (PHQ9) | -1.42 [-1.75 to -1.09]

6. Secondary Outcome: HIV Viral Control Change and Substance Use
Description: Change in participants with well controlled HIV RNA by 12 months after newly identified substance use problem
Time Frame: change between 24 months prior to clinic-specific implementation date and end of implementation period, up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation | Post-implementation (Clinical) | Post-implementation (Survey)
Number analyzed (Participants) | 974 | 189 | 580
Participants | 867 | 164 | 551

7. Secondary Outcome: HIV Viral Control Change and Mental Health
Description: Change in participants with well controlled HIV RNA by 12 months after newly identified mental health problem
Time Frame: change between 24 months prior to clinic-specific implementation date and end of implementation period, up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation | Post-implementation (Clinical) | Post-implementation (Survey)
Number analyzed (Participants) | 1088 | 261 | 269
Participants | 990 | 240 | 253

ADVERSE EVENTS:
Time Frame: Up to 3 years and 9 months (Up to 2 years pre-implementation + up to 21 months post-implementation)
Arm/Group | Pre-implementation | Post-implementation
All-Cause Mortality (participants affected / at risk) | 0/5706 | 0/5115
Serious Adverse Events (participants affected / at risk) | 0/5706 | 0/5115
Other Adverse Events (participants affected / at risk) | 0/5706 | 0/5115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03217058/Prot_000.pdf